CLINICAL TRIAL: NCT02527694
Title: Comparison of Quality of Cardiopulmonary Resuscitation Between Flexible Stretcher and Standard Stretcher in Out-of-Hospital Cardiac Arrest: Ambulance Stretcher Innovation of Asian CPR (ASIA-CPR) Trial
Brief Title: CPR Quality Between Flexible Stretcher and Standard Stretcher in OHCA
Acronym: ASIA-CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Do Shin, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-EM-2015-2P
Record Dates: First submitted 2015-08-06; First posted 2015-08-19 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2018-12

CONDITIONS: Out-of-hospital Cardiac Arrest
Keywords: Emergency medical services; Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flexible EMS Stretcher Cart Group (Experimental): Patients in this group will be transported on the new flexible EMS stretcher cart and receive mechanical CPR during transport to the hospital. The intervention will be given during elevator transport (if applicable) as well as in the moving ambulance.
  Interventions: Device: Flexible EMS stretcher cart; Device: mechanical CPR
- Standard Stretcher Cart Group (No Intervention): Patients in this group will be transported on the standard stretcher cart and receive manual CPR during transport to the hospital. The resuscitation protocol will follow the current standard protocol used by the EMS providers.

INTERVENTIONS:
Device: Flexible EMS stretcher cart — The flexible EMS stretcher cart is an innovative EMS stretcher cart built to be flexible to fit in smaller spaces such as elevators. The flexible stretcher bends at the hip joint as well as at the knee joint, so that the patient can be put in head-up position at 30 degrees elevation with elevated legs.
  Arms: Flexible EMS Stretcher Cart Group
Device: mechanical CPR
  Arms: Flexible EMS Stretcher Cart Group

SUMMARY:
This study aims to compare the quality of emergency medical services cardiopulmonary resuscitation between flexible stretcher and standard stretcher during ambulance transport to hospital among out-of-hospital cardiac arrest patients.

DETAILED DESCRIPTION:
Background: Cardiopulmonary resuscitation (CPR) during ambulance transport in Asia has been known to be ineffective for quality and unsafe for emergency medical services(EMS)providers. Small elevators in high rise buildings are the most serious barriers to provide high quality CPR due to too long stretcher cart to enter in the elevators. We developed flexible stretcher cart to be safely used in small elevator through reducing the length of the stretcher. This study aims to compare the quality of EMS CPR between flexible stretcher and standard stretcher during transport to hospital.

Method:

This is a before and after-trial in a metropolis EMS. Study targets are adult out-of-hospital cardiac arrest (OHCA), excluding evident death cases, pregnancy, DNR cases, and too big or too small body size for stretcher cart or mechanical CPR devices. In the before period, the standard stretcher will be used for manual CPR using standard CPR protocol. In the after period, the flexible stretcher will be used with mechanical CPR devices after 3 cycles of standard manual CPR. Individual and Utstein risk factors will be collected. Main outcomes are no-flow fraction (NFF) measured by defibrillators (X-series) and safety will be measured on mechanical error, transportation error, patient injury and EMS provider injury. Sample size were 24 cases for before (12 cases) and after (12 cases) trial from 80% power and 0.05 of alpha error for expecting 20% quality difference (30% NFF inflexible stretcher and 50% NFF in standard stretcher)

Expected impact:

The study will be expected to find the benefit of flexible stretcher cart during CPR in small elevators. This findings will contribute to revise the Asian EMS protocol for improving quality of CPR.

ELIGIBILITY:
Inclusion Criteria:

* All EMS-assessed OHCA in (3-4) selected districts in Seoul
* 18 years or older of age

Exclusion Criteria:

* Do-Not-Resuscitation cases or OHCA occurring in result of terminal diseases
* Signs of evident death (decapitation, evident livor mortis or rigor mortis)
* Pregnant
* Physique too large for mechanical CPR device application
* Chest deformation or injury
* EMS CPR quality not assessed by the defibrillator
* Return of spontaneous circulation (ROSC) before scene departure
* Cardiac arrest cases during transport

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Do Shin, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult OHCAs transported by five ambulances in a metropolitan area with a population of 3.5 million (many of whom lived in high-rise buildings) from September to October (before-phase) and November to December (afterphase) in 2015 were collected.
Groups:
- Flexible Stretcher Cart Group: Patients in this group will be transported on the new flexible stretcher cart and receive mechanical CPR during transport to the hospital. The intervention will be given during elevator transport (if applicable) as well as in the moving ambulance.
  Flexible EMS stretcher cart: The flexible stretcher cart is an innovative EMS stretcher cart built to be flexible to fit in smaller spaces such as elevators. The flexible stretcher bends at the hip joint as well as at the knee joint, so that the patient can be put in head-up position at 30 degrees elevation with elevated legs.
  mechanical CPR
Period: Overall Study
Arm/Group | Flexible Stretcher Cart Group | Standard Stretcher Cart Group
Started | 20 | 29
Completed | 10 | 21
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Population: During the before-phase, 29 OHCAs were treated and transported by EMS crews. After serial exclusion, 21 patients were eligible for the final analysis. During the afterphase, 20 OHCAs were eligible for enrollment. After serial exclusion, 10 cardiac arrests received mechanical chest compressions on reducible stretchers during hospital transport
Groups:
- Standard Stretcher Cart Group: Standard strecher for manual compression on supine position
- Flexible Stretcher Cart Group: We manufactured a stretcher that hinged at multiple points to be reduced to fit into small elevators with a patient on board. The stretcher can be used to transport patients without cardiac arrest in the same manner as a standard stretcher. In cases of cardiac arrest, the upper mattress of the stretcher could be removed to install the mechanical compression device. The stretcher has additional sidebars that can be used to attach and lock mechanical CPR devices that are commercially available in Korea. The patient' legs were elevated with V shape body position through knee flection and hip flection on accessory steel bar when the patients are being transporting to avoid decrease of venous return by leg-down. A l0ad-distributing band-type mechanical compression device, the AutoPulse® (ZOLL Medical, Chelmsford, MA, USA), was used for this study.
- Total: Total of all reporting groups
Arm/Group | Standard Stretcher Cart Group | Flexible Stretcher Cart Group | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 11 | 6 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 73] | 66 [60 to 74] | 66 [58 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 10
  Male | 13 | 8 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 21 | 10 | 31

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Percentage of Chest Compression Fraction Between Before- and After-phase Groups
Description: Chest compression fraction was calculated as proportion of CPR time spent providing compressions.
Time Frame: During the total prehospital resuscitation time
Measure: Median (Inter-Quartile Range); unit: Percentage of chest compression fraction
Arm/Group | Standard Stretcher Cart Group | Flexible Stretcher Cart Group
Number analyzed (Participants) | 21 | 10
Percentage of chest compression fraction | 80.1 [68.0 to 85.2] | 85.2 [83.4 to 86.3]

2. Secondary Outcome: CPR Duration
Time Frame: During total prehospital resuscitation
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Standard Stretcher Group: Standard strecher for manual compression on supine position
- Reducible Stretcher Group: We manufactured a stretcher that hinged at multiple points to be reduced to fit into small elevators with a patient on board. The stretcher can be used to transport patients without cardiac arrest in the same manner as a standard stretcher. In cases of cardiac arrest, the upper mattress of the stretcher could be removed to install the mechanical compression device. The stretcher has additional sidebars that can be used to attach and lock mechanical CPR devices that are commercially available in Korea. The patient' legs were elevated with V shape body position through knee flection and hip flection on accessory steel bar when the patients are being transporting to avoid decrease of venous return by leg-down. A l0ad-distributing band-type mechanical compression device, the AutoPulse® (ZOLL Medical, Chelmsford, MA, USA), was used for this study.
Arm/Group | Standard Stretcher Group | Reducible Stretcher Group
Number analyzed (Participants) | 21 | 10
seconds | 909 [594 to 1013] | 1131 [974 to 1262]

ADVERSE EVENTS:
Time Frame: During the 6 weeks of before-phase and 2 weeks of after-phase for a total of 2 months
Arm/Group | Standard Stretcher Group | Reducible Stretcher Group
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/20
Other Adverse Events (participants affected / at risk) | 0/29 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No